CLINICAL TRIAL: NCT01269788
Title: Comparing Omeprazole With Fluoxetine for Treatment of Non Erosive Reflux Disease and Its Subgroups: a Double-blind Placebo-controlled Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 89-02-30-10638
Record Dates: First submitted 2010-12-21; First posted 2011-01-04 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Non-erosive Reflux Disease
Keywords: non-erosive reflux disease; heartburn; functional; Antidepressive Agents, Second-Generation; Proton Pump Inhibitors
MeSH Terms: conditions — Non-Erosive Reflux Disease; Heartburn | interventions — Fluoxetine; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- pH positive-omeprazole (Active Comparator)
  Interventions: Drug: Omeprazole
- pH positive-placebo (Placebo Comparator)
  Interventions: Drug: placebo
- pH positive-fluoxetine (Active Comparator)
  Interventions: Drug: Fluoxetine
- pH negative-omeprazole (Active Comparator)
  Interventions: Drug: Omeprazole
- pH negative-fluoxetine (Active Comparator)
  Interventions: Drug: Fluoxetine
- pH negative-placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fluoxetine — 20 mg , oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH positive-fluoxetine
Drug: Omeprazole — 20 mg , oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH positive-omeprazole
Drug: placebo — oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH positive-placebo
Drug: Omeprazole — 20 mg , oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH negative-omeprazole
Drug: Fluoxetine — 20 mg , oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH negative-fluoxetine
Drug: placebo — oral , daily 30 mins before breakfast, for 6 weeks
  Arms: pH negative-placebo

SUMMARY:
Gastro-esophageal reflux disease (GERD) is highly prevalent, affecting up to 20% of the adult population in North America. Up to 70% of GERD patients have non-erosive reflux disease (NERD), a term used to describe symptoms suggestive of GERD in patients with no endoscopic evidence of erosive esophagitis. NERD represents a heterogeneous group of patients whom are sub classified according to 24 hours-PH monitoring results and also symptom-acid association analysis(Symptom Index,SI).

Treatment of NERD can be a challenge for clinicians. According to the many studies , the pooled rate for symptomatic response after a period of proton pomp inhibitor(PPIs)therapy as the most frequently used drug, in NERD patients is lower than for erosive esophagitis patients. It is also shown that acid exposure is much lower in NERD patients than those with erosive esophagitis and NERD patients are less likely to exhibit a strong association between heartburn symptoms and acid reflux events than patients with erosive oesophagitis.

Furthermore, beside the high economic burden, there are concerns about the adverse effects of long time administration of PPIs.

Several hypothesis has been proposed to describe low response rate of NERD patients to PPIs. One of the most acceptable theories is that patients with anxiety or depression and psychological problems are at an increased risk of developing reflux symptoms. On the other hand, pain modulators such as sertraline, a selective serotonin reuptake inhibitor(SSRI), and other antidepressants have been shown to improve symptoms in patients with functional gastrointestinal disorders like non cardiac chest pain.

According to the above-mentioned tips, the investigators hypothesize that antidepressants like fluoxetine, as an SSRI, may have beneficial effects in improving symptoms of NERD patients.

The purpose of this study is to compare the effect of omeprazole with fluoxetine and placebo for treatment of NERD patients and its subgroups who all experience reflux symptoms and have normal endoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 and below 60 years old
* experiencing heartburn during last 6 months before inclusion
* experiencing heartburn during at least 4 of 7 days before inclusion
* presence of normal mucosa in upper gastrointestinal(GI) endoscopy which has been documented during 7 days before inclusion provided that the patient has not administered any PPI during last 30 days before inclusion

Exclusion Criteria:

* inability to undergone upper GI endoscopy or PH monitoring
* presence of barret's esophagus or erosive esophagitis in upper GI endoscopy
* presence of active peptic ulcer disease or any disease which affects the absorption of drugs such as inflammatory bowel disease
* past history of esophageal or gastric surgery
* esophageal stricture which needs dilation
* administration of proton pomp inhibitors during 30 days before inclusion to the study
* administration of H2 blockers, anticholinergics, sucralfate and pro-kinetics during the assessments for eligibility and also during the study
* long time administration of non-steroidal anti-inflammatory drugs (NSAIDs)
* administration of neuroleptic or antidepressant drugs during 30 days before inclusion to the study
* known allergy to PPIs or SSRIs
* presence of significant systemic disease such as scleroderma , diabet mellitus , peripheral and autonomic neuropathies and ...
* pregnancy for females
* presence of known psychiatric disorder such as depression , panic disorder or drug addiction according to the DSM-IV criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
investigator-reported symptom severity | 6 weeks
  symptom severity at beginning and 6 weeks after the study ,assessed by the standard questionnaire

SECONDARY OUTCOMES:
patient-reported symptom severity | 6 weeks
  symptom severity reported by the patient in daily diary
heartburn-free days | 6 weeks
  percentage of 24-h heartburn-free days (days with neither daytime nor nighttime heartburn) during treatment assessed by daily diary

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Amir Mirbagheri, MD, Study Chair — Department of Internal Medicine, Faculty of medicine, Tehran university of medical sciences; Mohammad Reza Ostovaneh, MD,MPH, Principal Investigator — Tehran University of Medical Sciences; Arash Etemadi, MD, PhD, Principal Investigator — Tehran University of Medical Sciences; Yasin Farrokhi Khajeh Pasha, MD, MPH, Principal Investigator — Tehran University of Medical Sciences; Behtash Saeidi, MD, Principal Investigator — Tehran University of Medical Sciences; Kaveh Hajifathalian, MD, Principal Investigator — Tehran University of Medical Sciences; Akbar Fotouhi, MD, PhD, Principal Investigator — Tehran University of Medical Sciences; Seyed Mahmoud Eshagh hosseini, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gasterointestinal endoscopy ward, Amir Alam hospital, Tehran university of medical sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Heidelbaugh JJ, Goldberg KL, Inadomi JM. Overutilization of proton pump inhibitors: a review of cost-effectiveness and risk [corrected]. Am J Gastroenterol. 2009 Mar;104 Suppl 2:S27-32. doi: 10.1038/ajg.2009.49. PMID 19262544
- [Background] Martinez SD, Malagon IB, Garewal HS, Cui H, Fass R. Non-erosive reflux disease (NERD)--acid reflux and symptom patterns. Aliment Pharmacol Ther. 2003 Feb 15;17(4):537-45. doi: 10.1046/j.1365-2036.2003.01423.x. PMID 12622762
- [Background] Raghunath AS, O'Morain C, McLoughlin RC. Review article: the long-term use of proton-pump inhibitors. Aliment Pharmacol Ther. 2005 Aug;22 Suppl 1:55-63. doi: 10.1111/j.1365-2036.2005.02611.x. PMID 16042660
- [Background] Dean BB, Gano AD Jr, Knight K, Ofman JJ, Fass R. Effectiveness of proton pump inhibitors in nonerosive reflux disease. Clin Gastroenterol Hepatol. 2004 Aug;2(8):656-64. doi: 10.1016/s1542-3565(04)00288-5. PMID 15290657
- [Background] Bradley LA, Richter JE, Pulliam TJ, Haile JM, Scarinci IC, Schan CA, Dalton CB, Salley AN. The relationship between stress and symptoms of gastroesophageal reflux: the influence of psychological factors. Am J Gastroenterol. 1993 Jan;88(1):11-9. PMID 8420248
- [Background] DeVault KR. Review article: the role of acid suppression in patients with non-erosive reflux disease or functional heartburn. Aliment Pharmacol Ther. 2006 Mar;23 Suppl 1:33-9. doi: 10.1111/j.1365-2036.2006.02798.x. PMID 16483268
- [Background] Venes DJ. Imipramine in patients with chest pain despite normal coronary angiograms. N Engl J Med. 1994 Sep 29;331(13):882; author reply 882-3. No abstract available. PMID 8078547
- [Background] Handa M, Mine K, Yamamoto H, Hayashi H, Tsuchida O, Kanazawa F, Kubo C. Antidepressant treatment of patients with diffuse esophageal spasm: a psychosomatic approach. J Clin Gastroenterol. 1999 Apr;28(3):228-32. doi: 10.1097/00004836-199904000-00008. PMID 10192608
- [Background] Varia I, Logue E, O'connor C, Newby K, Wagner HR, Davenport C, Rathey K, Krishnan KR. Randomized trial of sertraline in patients with unexplained chest pain of noncardiac origin. Am Heart J. 2000 Sep;140(3):367-72. doi: 10.1067/mhj.2000.108514. PMID 10966532
- [Background] Broekaert D, Fischler B, Sifrim D, Janssens J, Tack J. Influence of citalopram, a selective serotonin reuptake inhibitor, on oesophageal hypersensitivity: a double-blind, placebo-controlled study. Aliment Pharmacol Ther. 2006 Feb 1;23(3):365-70. doi: 10.1111/j.1365-2036.2006.02772.x. PMID 16422995
- [Background] Rentz AM, Kahrilas P, Stanghellini V, Tack J, Talley NJ, de la Loge C, Trudeau E, Dubois D, Revicki DA. Development and psychometric evaluation of the patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) in patients with upper gastrointestinal disorders. Qual Life Res. 2004 Dec;13(10):1737-49. doi: 10.1007/s11136-004-9567-x. PMID 15651544
- [Background] Fass R, Chey WD, Zakko SF, Andhivarothai N, Palmer RN, Perez MC, Atkinson SN. Clinical trial: the effects of the proton pump inhibitor dexlansoprazole MR on daytime and nighttime heartburn in patients with non-erosive reflux disease. Aliment Pharmacol Ther. 2009 Jun 15;29(12):1261-72. doi: 10.1111/j.1365-2036.2009.04013.x. Epub 2009 Apr 8. PMID 19392864
- [Derived] Ostovaneh MR, Saeidi B, Hajifathalian K, Farrokhi-Khajeh-Pasha Y, Fotouhi A, Mirbagheri SS, Emami H, Barzin G, Mirbagheri SA. Comparing omeprazole with fluoxetine for treatment of patients with heartburn and normal endoscopy who failed once daily proton pump inhibitors: double-blind placebo-controlled trial. Neurogastroenterol Motil. 2014 May;26(5):670-8. doi: 10.1111/nmo.12313. Epub 2014 Feb 7. PMID 24533896